CLINICAL TRIAL: NCT05921474
Title: Detection of Circulating Tumor DNA After Stereotactic Ablative Radiotherapy in Patients With Unbiopsied Lung Tumors
Acronym: SABR-DETECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: SABR-DETECT
Record Dates: First submitted 2023-02-15; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Early Stage Lung Cancer; Stage I/IIA; Tumor stage T1-T2b
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma will be collected for circulating tumor DNA (ctDNA) and cancer detection analysis at eight time-points. At each time-point, four 10 mL [Paxgene circulating cell-free DNA (ccfDNA), Streck blood collection tube (BCT) or K2EDTA] tubes will be drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Unbiopsied, Presumed Stage I/IIA NSCLC Undergoing SABR: The first cohort will be comprised of patients with suspected stage I/IIA NSCLC with plans to undergo curative SABR.
- Patients with Stage I-IIA NSCLC Undergoing SABR: The second cohort will be comprised of patients with biopsy proven NSCLC, with clinically staged I/IIA disease with a plan to undergo definitive therapy with SABR.

SUMMARY:
The goal of this observational study is to determine if liquid biopsies from patients with stage I non-small cell lung cancer (NSCLC) can add to the diagnosis of a small lung cancer, or can better detect recurrent lung cancer compared to the standard of care procedures used for diagnosing this type of cancer. The main question[s] it aims to answer are:

* Primary Objective:

  1) To assess whether liquid biopsy for molecular residual disease during follow-up can predict a recurrence of lung cancer
* Secondary Objectives:

  1. To assess the impact of SABR on detection rates of ctDNA in patients undergoing SABR for early-stage lung tumors.
  2. To correlate positivity by blood-based cancer detection platforms and pre-treatment probability of malignancy using the Brock and Herder models.

Study investigators will also assess the rate of detection for targetable mutations in this patient population, and to correlate ctDNA findings, in patients without tissue confirmed disease.

Blood samples from participants will collected at eight (8) time-points: before the participant's first radiation treatment, following their first treatment and then at their 3-month, 6-month, 9-month, 12-month, 18-month and 24-month follow-up visits.

DETAILED DESCRIPTION:
This is a multi-institutional cohort study. The first cohort will be comprised of patients with suspected stage I/IIA NSCLC with plans to undergo curative SABR. The second cohort will be comprised of patients with biopsy proven NSCLC, with clinically staged I/IIA disease with a plan to undergo definitive therapy with SABR.

Focused, or stereotactic, radiation therapy is a standard treatment for early-stage lung cancer when surgery is not possible due to comorbidities or when patient denies surgery and opts for radiation therapy. Many patients with early stage (1 or 2) disease often have treatment with radiation without a tissue biopsy, because of the risk associated with the procedure of tissue biopsy. If the chances of mass being spread to other organs are very high, the risk of treating a lesion with radiation without a biopsy is less than the risk of a biopsy. Unfortunately, many of these patients will have their cancer come back at the local site or at a new site (10-20% risk of recurrence at 1 year). At such time they need a tissue biopsy for diagnosis and biomarker testing to decide the best treatment options. The time to get a biopsy and complete results can take over a month.

Liquid biopsy is a type of test which isolates the cancer derived circulating DNA from blood. This DNA can be tested for mutations and other changes. This offers a chance to diagnose cancer patients in whom biopsy is not possible, or may provide the result faster or safer than a conventional biopsy. Additionally, liquid biopsies can detect mutations which can be used to guide treatment if cancer comes back (recurs); and treatment could be started without a biopsy or immediately after the biopsy before the results are available. It may also help detect a recurrence earlier compared to surveillance imaging.

This study, SABR-DETECT may answer these questions -

1. Can the investigators detect a recurrence earlier with a liquid biopsy, compared to standard surveillance with CT scans?
2. Can radiation increase the ability to diagnose cancer when the baseline liquid biopsy test is negative?
3. Can liquid biopsy be used for diagnosis of lung cancer in patients when a tissue biopsy is not possible or the risks are too high?

Plasma will be collected for ctDNA and cancer detection analysis at eight time-points. At each time-point, four 10 mL (Paxgene ccfDNA, Streck BCT or K2EDTA) tubes will be drawn.

* Draw #1: prior to the first fraction of SABR, ideally on the same day as treatment (but before treatment delivery).
* Draw #2: this should be collected on the second day after the first fraction (± 24 hours if collection is not feasible on that day). For example, if the first treatment is on a Monday, the second collection should occur on a Wednesday, but may occur anytime between Tuesday and Thursday.
* Draws #3-8: at 3-month, 6-month, 9-month, 12-month, 18-month and 24-month follow-up, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Willing to provide informed consent
* Undergoing SABR for a solitary pulmonary nodule (SPN) with tissue confirmation or those without tissue confirmation of malignancy, must have a pretreatment likelihood of malignancy of ≥ 60% using either the Herder or Brock models (60% probability was chosen to have a reasonable chance that there will indeed be cancer in the nodule; however, most patients are expected to have a pretreatment probability of > 85%).
* Tumor stage T1-T2b (≤ 5 cm)
* No evidence of nodal or distant metastases
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3

Exclusion Criteria:

* Contraindications to radiotherapy
* Prior history of any invasive malignancy within 5 years, which might interfere with the interpretation of the ctDNA results. Non-melanoma skin cancer is allowed if under appropriate control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Stage I/IIA Non-small cell lung cancer that will undergo Stereotactic Ablative Radiotherapy (SABR) for a solitary pulmonary nodule with tissue confirmation or those without tissue confirmation of malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To assess whether liquid biopsy for molecular residual disease during follow-up can predict a recurrence of lung cancer. | End of study (approximately Dec 2023)
  Percentage of patients with MRD detected prior to or at the time of radiological recurrence, with longitudinal monitoring of ctDNA

SECONDARY OUTCOMES:
To assess the impact of SABR on detection rates of ctDNA in patients undergoing SABR for early-stage lung tumors. | End of study (approximately Dec 2023)
  * The percentage of patients with undetectable ctDNA at baseline who then develop detectable ctDNA after one fraction of SABR.
  * Increase in variant allelic frequency (vAF) or quantifiable ctDNA (mutant molecules/mL of plasma) from baseline to post-treatment samples, in patients with detectable ctDNA at baseline.
To correlate positivity by blood-based cancer detection platforms and pre-treatment probability of malignancy using the Brock and Herder models. | End of study (approximately Dec 2023)
  Correlation between pre-treatment malignancy risk to the rate of ctDNA positivity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Breadner, MD, Principal Investigator — 519-685-8640
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma S, Young S, Kennedy TAC, Carvalhana I, Black M, Baer K, Churchman E, Warner A, Allan AL, Izaguirre-Carbonell J, Dhani H, Louie AV, Palma DA, Breadner DA. Detection of Circulating Tumor DNA After Stereotactic Ablative Radiotherapy in Patients With Unbiopsied Lung Tumors (SABR-DETECT). Clin Lung Cancer. 2024 Mar;25(2):e87-e91. doi: 10.1016/j.cllc.2023.11.013. Epub 2023 Dec 1. PMID 38101984